CLINICAL TRIAL: NCT06727786
Title: Using a Serious Game to Teach People How to Recognize and Respond to Opioid Overdose
Brief Title: Serious Game to Teach Opioid Overdose Response
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2159620
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention/training
- Serious Game (Experimental): Serious Game training to respond to opioid overdose
  Interventions: Other: Serious game training

INTERVENTIONS:
Other: Serious game training — A serious game featuring a dramatic/realistic film, pauses with questions for active learning, and practice administration of naloxone and performing CPR
  Arms: Serious Game

SUMMARY:
This study evaluates the efficacy of a serious game to teach students how to recognize and respond to opioid overdose

DETAILED DESCRIPTION:
This study uses an interactive realistic film depicting an opioid overdose to teach high school/middle school students how to recognize and respond to opioid overdose. The film features a person who finds their friend unresponsive, with evidence of opioid use. The unresponsive friend demonstrates signs of opioid overdose. The hero must recognize opioid overdose, administer naloxone (opioid antedote) and perform CPR. The film is made interactive by the narrator pausing the action of the film, and asking learners to answer questions/make choices.

Efficacy is tested on the day of training, and 2-4 months later. Efficacy is measured by student ability to correctly administer naloxone to a manikin, perform CPR, and answer knowledge questions about opioid overdose. Other studied metrics include student engagement/enjoyment, attitudes/biases, and emotions created by the training. These will be tested through validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Student at participating school, enrolled in Health or Science Class

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Naloxone administration Skill | Day of training, and 2-3 months
  Properly administer naloxone to a victim of opioid overdose Study personnel will ask students to administer naloxone to a CPR manikin. Personnel will use a checklist from the Center for Addiction and Mental Health to score student responses.

SECONDARY OUTCOMES:
CPR Skill | Day of training, and 2-3 months
  Ability to perform high-quality CPR Students will be asked to perform CPR on a CPR manikin for 2 minutes. CPR skill will be measured with the CPR Meter 2 from Laerdal, which reports compression rate, depth, and percent recoil. We will consider "high quality CPR" students who perform 70% or more of compressions at appropriate rate (100-120/min), depth (2-2.5inches), and full recoil.
Attitudes towards opioid overdose | Day of training, and 2-3 months
  Attitudes, enjoyment, and emotions towards opioid overdose
  Emotions will be measured using the PANAS scale (Positive And Negative Affect Scale) which consists of 10 positive and 10 negative emotion words. The total score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect.
  Engagement and enjoyment will be measured using Likert-style questions asking for agreement with statements such as "I enjoyed CPR training," "CPR training was fun," "I will use CPR training in the future," "It is important to learn CPR"
  Attitudes will be measured with a custom questionnaire asking Likert-style responses to statements regarding opioid overdose.
Knowledge of opioid overdose response | Day of training, and 2-3 months
  Knowledge of how to recognize and respond to opioid overdose A questionnaire of custom-created multiple choice questions will assess student knowledge of how to recognize and respond to opioid overdose.

IPD SHARING:
Plan to Share IPD: No
Participants are minors and therefore protected. No IDP will be shared